CLINICAL TRIAL: NCT02057913
Title: A Phase II Trial of Vinflunine Chemotherapy in Locally-advanced and Metastatic Carcinoma of the Penis
Brief Title: A Phase II Trial of Vinflunine Chemotherapy in Locally-advanced and Metastatic Carcinoma of the Penis (VinCaP)
Acronym: VinCaP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institute of Cancer Research, United Kingdom (Other)
Collaborators: St George's Healthcare NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ICR-CTSU/2012/10036; CRUK/12/021 (Other Grant/Funding Number: Cancer Research UK); 2012-002592-34 (EudraCT Number); 13/LO/0822 (Other: Main REC number); CCR3858 (Other: Sponsor Number)
Record Dates: First submitted 2014-02-05; First posted 2014-02-07 (Estimated); Last update posted 2020-07-23 (Actual); Status verified 2018-08

CONDITIONS: Locally-advanced or Metastatic Penile Neoplasms
Keywords: Penile neoplasms; Chemotherapy; Vinflunine; Phase II
MeSH Terms: conditions — Penile Neoplasms | interventions — vinflunine

ARMS (1):
- Vinflunine (Experimental): All patients will receive on Day 1 of a 21 day cycle, vinflunine 320mg/m2 via intravenous infusion in either 100ml sodium chloride 0.9% or glucose 5% over 20 minutes; four cycles to be given in total prior to formal re-staging.
  Interventions: Drug: Vinflunine

INTERVENTIONS:
Drug: Vinflunine — All patients will receive on Day 1 of a 21 day cycle, vinflunine 320mg/m2 via intravenous infusion in either 100ml sodium chloride 0.9% or glucose 5% over 20 minutes; four cycles to be given in total prior to formal re-staging.
  Other Names: Javlor

SUMMARY:
VinCaP is a multicentre single-arm phase II trial. 22 patients will receive Vinflunine chemotherapy (Vinflunine 320mg/m2 given intravenously on day 1 of each cycle of 21 days, four cycles to be given prior to formal re-staging).

ELIGIBILITY:
Inclusion Criteria:

1. Male, ≥18 years.
2. Measurable disease as determined by RECIST (Response Evaluation Criteria in Solid Tumors) criteria (version 1.1).
3. Patients who present with purely cutaneous measurable disease should fulfill RECIST Criteria (see Appendix 1). Lesions should be a minimum size of 10 mm and measured using calipers by clinical examination.
4. Histologically-proven squamous cell carcinoma of the penis.
5. Stage: M1, or; M0, any T, N3 (i.e. involvement of deep inguinal or pelvic lymph nodes) or; M0, any T, N2 (i.e. involvement of multiple or bilateral superficial lymph nodes) or; M0, T4 (tumour invades other adjacent structures) any N.

   Notes:
   1. Patients with M0 disease may be considered if, in the opinion of the specialist Multi Disciplinary Team (MDT), they are deemed unlikely to benefit from surgery with curative intent and unlikely to tolerate combination chemotherapy due to comorbidities and/or disease burden.
   2. Patients who have received prior radiotherapy to non-target lesions may be included.
6. Pre-treatment blood counts, haematology and biochemistry values within the following acceptable limits: Absolute Neutrophil Count (ANC) ≥ 1,500/mm3, Platelets ≥100,000/mm3, glomerular filtration rate (GFR) ≥60ml/min. GFR to be assessed according to local practice (recommended technique of eGFR using the MDRD formula.
7. Liver function: Patients must have (with or without the presence of liver metastases):

   * A prothrombin time >70% normal value (NV) AND
   * Bilirubin <1.5xUpper Limit of Normal (ULN) AND
   * Transaminases <2.5xULN AND
   * GGT <5xULN
8. Performance Status Eastern Cooperative Oncology Group (ECOG) 0, 1 or 2.
9. Written, informed consent.

Exclusion Criteria:

1. Pure verrucous carcinoma of the penis.
2. Squamous carcinoma of the urethra.
3. Patients who do not have measurable disease as determined by RECIST (version 1.1).
4. T1 N1 M0 disease.
5. T2 N1 M0 disease.
6. M0, T3, N1 (tumour invades urethra or prostate and single inguinal node involved).
7. Unfit for vinflunine chemotherapy (as assessed by the multidisciplinary team).
8. Previous chemotherapy or chemoradiotherapy.
9. Contraindication to chemotherapy.
10. Other malignancy (other than Squamous Cell Carcinoma or Basal Cell Carcinoma of non-penile skin) that has required surgical or non-surgical treatment in the last 5 years. All patients with a previous cancer diagnosis must be discussed the Chief Investigator prior to entry into the trial.
11. Patients who have received radiotherapy to target lesions and have no other lesions that can act as target lesions instead:

    e.g. Patients with recurrent pelvic lymph nodes that are deemed irresectable and who have had prior radiotherapy to those lymph nodes:

    i. are INELIGIBLE if the involved lymph nodes are the only site of disease.

    ii. are ELIGIBLE if they have other measurable sites of disease e.g. pulmonary metastases.

    If uncertain, please discuss with the Chief Investigator.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2014-03-17 (Actual); Primary Completion 2018-11-06 (Actual); Study Completion 2018-11-06 (Actual)

PRIMARY OUTCOMES:
Clinical Benefit | 12 weeks
  To determine the clinical benefit (objective response & stable disease rate) and toxicity of vinflunine in patients with inoperable (locally advanced or metastatic) cancer of the penis and thus determine whether this drug warrants further research in this indication.

SECONDARY OUTCOMES:
Objective Response Rate | 12 weeks
  Proportion of patients having achieved partial or complete remission. The proportion of patients with objective response will be calculated and presented along its 95% confidence interval.
Toxicity | Baseline, 3, 6, 9, 12 weeks on treatment, and at follow-up, 3, 6, 9, 12, 18, 24 months (timed from end of last cycle of chemotherapy)
  Toxicity will be evaluated, using the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) v4 scoring, after each cycle, at the end of treatment and at follow up visits. The proportion of patients experiencing grade 3 or 4 toxicities at these time points and until progression will be reported as well as the Serious Adverse Events (SAEs).
Progression-free survival | From registration to first documented disease progression or death from any cause, up to 24 months
  Progression-free survival will be defined as time from registration until the first of clinically or radiologically documented disease progression, or death from any cause death. Patients alive and progression-free at time of analysis will be censored at date last seen.
Overall Survival | Time from registration until death from any cause, up to 24 months
  Patients alive at time of analysis will be censored at date last seen. Patients lost to follow-up will be censored at date last seen.
Treatment Compliance | 12 weeks
  Treatment Compliance will be defined as proportion of planned doses delivered. Reasons for non-delivery of planned doses (patient or clinician preference, toxicity and tolerability) will be collected.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Pickering, MBBS, MRCP, Principal Investigator — St George's Healthcare NHS Trust
Locations (9):
- United Kingdom (9):
  - Velindre NHS Trust, Whitchurch, Cardiff
  - Royal Cornwall Hospitals NHS Trust, Truro, Cornwall
  - University College London Hospitals NHS Foundation Trust, London, Greater London
  - The Christie NHS Foundation Trust, Manchester, Greater Manchester
  - St George's Healthcare NHS Trust, Tooting, London
  - Clatterbridge Centre for Oncology NHS Foundation Trust, Metropolitan Borough of Wirral, Merseyside
  - Beatson West of Scotland Cancer Centre, Glasgow
  - St James's University Hospital, Leeds
  - Leicester Royal Infirmary, Leicester

REFERENCES:
- [Derived] Nicholson S, Tovey H, Elliott T, Burnett SM, Cruickshank C, Bahl A, Kirkbride P, Mitra AV, Thomson AH, Vasudev N, Venugopal B, Slade R, Tregellas L, Morgan B, Hassall A, Hall E, Pickering LM. VinCaP: a phase II trial of vinflunine in locally advanced and metastatic squamous carcinoma of the penis. Br J Cancer. 2022 Jan;126(1):34-41. doi: 10.1038/s41416-021-01574-9. Epub 2021 Oct 20. PMID 34671131